CLINICAL TRIAL: NCT05768074
Title: Family Therapy Training and Implementation Platform (FTTIP): An Innovative Web-based Tool for Long-term Practice Improvement Supplement Study
Brief Title: Family Therapy Training and Implementation Platform (FTTIP) Supplement Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Training and Implementation Associates (Other)
Responsible Party: Sponsor
Other Study IDs: 3R44MH115547-02S1 (NIH)
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Traditional Face to Face Training; Family Therapy Training and Implementation Platform (FTTIP)
Keywords: Mental health; Family therapy; Mental health training
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Therapists: 20 therapists who were already trained will participate in a qualitative interview to gather perceptions and experiences of the therapists about the process of learning and practicing specific CIFFTA competencies from the therapy training platform (time 1 interview) and later, about their unique experiences related to implementation of the Evidenced Based Treatment (EBT), delivery of competencies learned, and the application of EBT in a real-world context (time 2).
  Interventions: Other: Qualitative Interview
- Agency leaders: 16 agency leaders from the main study will participate in qualitative interviews to 2) gain a deeper understanding from leaders of their experiences in facilitating EBTs at their agencies, the identification of barriers that can be addressed by the organizational readiness work (time 1), and later regarding their agencies experience with the platform, consultation process, perceived cost-benefit, and agency readiness (at time 2).
  Interventions: Other: Qualitative Interview

INTERVENTIONS:
Other: Qualitative Interview — Therapists and agency leaders receiving intervention from the main study will participate in qualitative interviews

SUMMARY:
The goal of this observational study is to learn about therapists' and agency leaders' experience with evidenced based treatments and the Family Therapy Training and Implementation Platform (FTTIP).

The main questions it aims to answer are:

1. What are the perceptions and experiences of the therapists about the process of learning and practicing specific Culturally Informed Flexible Family Based Treatment for Adolescents (CIFFTA) competencies from the platform?
2. What are therapists' unique experiences related to implementation of the evidenced based treatment (EBT), delivery of competencies learned, and the application of EBT in a real-world context?
3. What are agency leaders' experiences in facilitating EBTs at their agencies what are the barriers that can be addressed by the organizational readiness work?
4. What is the experience of the entire agency with the platform, consultation process, perceived cost-benefit, and agency readiness?

DETAILED DESCRIPTION:
The supplement project will have multiple components that augment the parent study by collecting qualitative data that we can combine with the parent study's quantitative data to better understand the experiences of trainees and agency leaders with the platform.Twenty trainees (randomly selected from the 75 CIFFTA parent study trainees) and 16 agency leaders from the sample of the parent study will be included. The proposed supplement aims to: 1) gather perceptions and experiences of the trainees about the process of learning and practicing specific CIFFTA competencies from the platform (time 1 interview) and later, about their unique experiences related to implementation of the EBT, delivery of competencies learned, and the application of EBT in a real-world context (time 2); and 2) gain a deeper understanding from leaders of their experiences in facilitating EBTs at their agencies, the identification of barriers that can be addressed by the organizational readiness work (time 1), and later regarding their agencies experience with the platform, consultation process, perceived cost-benefit, and agency readiness (at time 2).

ELIGIBILITY:
Inclusion Criteria:

* Bachelors level counselor with 2 years of experience or Master's level counselors and therapists who have not had family therapy training in the past year and who are broadly representative of the potential trainees in the general population, including educational background and job experience with different client populations (e.g., varied demographics and presenting problems).
* All therapists must be actively providing treatment to youth and be willing to deliver the family intervention to at least one family during the project period
* Therapists must be enrolled in the parent grant and be randomized to the FTTIP condition
* Agency leaders must be enrolled in the parent grant study
* To be included in the study, agency leaders must have the authority to allocate agency resources (e.g., giving trainees protected time to participate in training activities, allowing smaller caseloads as they begin implementation) and be willing to participate in agency readiness and implementation consultation.

Exclusion Criteria:

* • We are not limiting inclusion of any group by sex/gender, race, and/or ethnicity

  * Agencies that are unwilling to participate in all study activities, that have nontraditional funding sources (e.g., totally charity funded), or that are so small they cannot assign sufficient counselors to the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be selected from therapists and agency leaders that are already enrolled in the parent study (150 counselors and 30 agency leaders).
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
TIA Therapist Interview Timepoint 1 | After 2 weeks given to complete a 20 hour training
  Interview to assess perceptions and experiences of the therapists about the process of learning and practicing specific CIFFTA competencies from the platform
TIA Therapist Interview Timepoint 2 | After four months of the implementation of the treatment with a family
  Interview to assess therapists' unique experiences related to implementation of the Evidenced Based Treatment, delivery of competencies learned, and the application of EBT in a real-world context
TIA Agency leader Interview Timepoint 1 | Prior to the start of training or implementation of therapists at the organization
  Interview to gain a deeper understanding from leaders of their experiences in facilitating EBTs at their agencies, the identification of barriers that can be addressed by the organizational readiness work
TIA Agency leader Interview Timepoint 2 | After four months of treatment implementation at the organization
  Interview to assess agencies experience with the platform, consultation process, perceived cost-benefit, and agency readiness

IPD SHARING:
Plan to Share IPD: No